CLINICAL TRIAL: NCT02897154
Title: Clinical Evaluation of i-STAT Analyzer for Glucose, Hematocrit and Sodium
Brief Title: Clinical Evaluation of i-STAT Analyzer Glucose, Hematocrit and Sodium for Capillary Samples
Status: Completed | Type: Observational
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-2016-0003
Record Dates: First submitted 2016-07-06; First posted 2016-09-13 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Analytical Performance of Sodium, Glucose and Hematocrit Assays by the i-STAT 500 (Alinity) Analyzer
MeSH Terms: interventions — In Vitro Meat

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: In-vitro

SUMMARY:
The objective of this study is to compare the performance of two i-STAT Analyzers in a Point-of-Care (POC) setting. The evaluation will be performed using a cartridge to test glucose, hematocrit and sodium on capillary specimens.

DETAILED DESCRIPTION:
The clinical performance for glucose, hematocrit and sodium assays for capillary samples was evaluated for the investigational i-STAT 500 (Alinity) analyzer based on results of method comparison testing against the i-STAT 1W analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subjects (or their legal representative) who are willing to voluntarily consent to the study

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (18 years or older)
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Glucose (mg/dL) levels | Patient's blood is tested within 3 minutes of blood collection
  Data analysis
Hematocrit (%PCV) levels | Patient's blood is tested within 3 minutes of blood collection
  Data analysis
Sodium (mmol/L) levels | Patient's blood is tested within 3 minutes of blood collection
  Data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Edwards, BSc, Study Director — Abbott Point of Care
Locations (3):
- United States (3):
  - Diablo Clinical Research, Walnut Creek, California
  - Kentucky Clinical Trials Laboratory, Louisville, Kentucky
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT02897154/SAP_000.pdf
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT02897154/Prot_001.pdf